CLINICAL TRIAL: NCT06861153
Title: Pulses: Optimizing Pulse Consumption for Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004194
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular (CV) Risk; Healthy Eating Index; HbA1c; Lipid Profile; CRP
Keywords: pulses; pulse consumption; cardiometabolic health; dietary intervention; nutrition education; chronic disease prevention; healthy eating; dietary guidelines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pulses 1.5 cups Group (Experimental): Participants will be prescribed a diet that integrates 1.5 cup-equivalents of pulses per week.
  They will receive tailored nutrition education, including one-on-one sessions with nutrition educators, focused on how to incorporate pulses into everyday meals.
  Biweekly cooking classes and food demonstrations will be provided to illustrate easy pulse-based recipes and methods of preparation.
  Interventions: Behavioral: Pulses 1.5 cups Group
- Pulses 3 cups Group (Experimental): Participants will receive an increased dose of 3 cup-equivalents of pulses per week.
  Similar to the first arm, they will participate in personalized nutrition education sessions and attend biweekly cooking classes and food demonstrations, all specifically designed to support a higher intake of pulses.
  Interventions: Behavioral: Pulses 3 cups Group
- My Plate Group (Control) (Active Comparator): Participants will continue with their habitual dietary practices without any prescribed increase in pulse consumption.
  This arm will receive general nutrition education sessions covering balanced dietary practices, but without any additional focus on pulse integration.

INTERVENTIONS:
Behavioral: Pulses 1.5 cups Group — Participants will receive 1.5 cup-equivalents of pulses per week.
  Arms: Pulses 1.5 cups Group
Behavioral: Pulses 3 cups Group — Participants will receive 3 cup-equivalents of pulses per week.
  Arms: Pulses 3 cups Group
Behavioral: My Plate Group (Control) — Participants will continue with their usual dietary practices, receiving no additional pulses. They are encouraged to follow My Plate general recommendations.

SUMMARY:
This randomized clinical trial aims to evaluate the effects of consuming two different doses of pulses (1.5 cups/week or 3 cups/week) in individuals with baseline intake below 1.5 cups/week, compared to a control group receiving standard nutrition education based on the United States Department of Agriculture's (USDA) My Plate guidelines.

The main question the Pulses study aims to answer is:

• What is the effect of increasing pulse consumption (in a dose-response manner) on specific cardiometabolic risk factors, including LDL-C, CRP, HBA1C, and blood pressure compared to standard nutrition education?

For secondary outcomes, this study aims to answer the following:

• Does increased pulse consumption improve the following: overall serum lipid profile (Total cholesterol (TC), HDL-C, Triglycerides (TG), diet quality (measured by the Healthy Eating Index), and participants self-reported satisfaction with life (SWLS) and Satisfaction with Food-related Life (SWFoL).

All participants will attend biweekly classes and food demonstrations. The pulses groups will learn to prepare various pulse-based recipes, while the control group will receive guidance on preparing healthy meals following the USDA MyPlate recommendations.

DETAILED DESCRIPTION:
This is a randomized, parallel-arm study with 3 groups: 1) Control (Con). This group will receive educational materials and attend a series of 6 cooking classes focused on the USDA's MyPlate guidelines; 2) Pulses 1.5. This group receive nutrition education and attend a series of 6 cooking classes focused on both USDA's MyPlate guidelines, with a specific emphasis on how to incorporate more pulses into their diet. They will also receive 1.5 cup-equivalents of pulses per week for 6 weeks to take home with them to prepare and eat; 3) Pulses 3.0.

This group will receive the same nutrition education and cooking classes as the Pulses1.5 group, but will be provided with 3.0 cup equivalents of pulses to prepare and eat per week. Participants will be randomized after baseline testing. RedCap will be used to randomly assign participants to a treatment sequence. The randomization ratio will be balanced (balanced by gender and number of participants in each group). Intervention periods must be at least 12 weeks, however participants may continue the intervention for up to 14 weeks total (as is indicated in the informed consent). The range of 12-14 weeks is designed to accommodate for scheduling challenges that may occur due to illness, travel, etc. For example, if a participant completes 12 weeks of the intervention but then is unable to come in for an endpoint visit immediately, we will be able to continue the intervention until they are available for testing. The 12-14 week range will help to accommodate for these scheduling requirements.

Screening: Participants will be screened via an online REDCap survey including demographic and eligibility questions. Individuals who qualify for participation in the study will be invited to schedule a baseline testing visit in our nutrition research center.

Baseline and Week-12 Visits: At the baseline visit, participants will sign an IRB-approved informed consent form. At both visits, following an overnight fast, a blood draw will be completed, and height, weight, and vital signs will be determined. Premenopausal women will be asked to come in for endpoint visits at same point in their menstrual cycle (within the same 5-7 day window) as their baseline visit. In addition, participants will complete questionnaires to assess satisfaction with life and their diet.

* Blood Sampling: A fasting blood draw will be performed at each assessment to measure biomarkers of cardiometabolic health (including but not limited to): total cholesterol (TC), triglycerides (TG), HDL-C, LDL-C, HbA1c, and CRP. Values will be determined according to standardized procedures via Quest Diagnostics.
* Blood Pressure: Brachial blood pressure (BP) will be assessed under standardized conditions using an automated cuff. The BP measurements will be taken following the Joint National Committee 7 (JNC7) blood pressure guidelines in a quiet, temperature-controlled, dimly lit room following a 5-minute seated rest period, asking them not to use their phones, not to talk, and not to cross their legs. 3 measurements will be made, with 30 seconds rest in between, and the average will be calculated.

Questionnaires:

* Satisfaction with Food-related Life (SWFoL) scale: This scale consists of five items, grouped into a single dimension, that evaluate a person's overall assessment of their food and eating habits (e.g., "Food and meals bring great satisfaction to my daily life").
* Satisfaction with Life Scale (SWLS): This scale consists of five items, grouped into a single dimension, which evaluate overall cognitive judgments about a person's own life (e.g., "In most ways my life is close to my ideal").
* International Physical Activity Questionnaire (IPAQ): This questionnaire assesses the amount of time spent being physically active during the last seven days, grouped into vigorous, moderate, walking, and sitting categories.

Dietary Assessment: At baseline, participants will be instructed to maintain their regular caloric intake. At both baseline and at 12 weeks, participants will complete a 3 day dietary record to assess their dietary intake. At each timepoint (baseline and 12 weeks), dietary records will be conducted on 3 separate days to capture their average intake over a week. Baseline 3-day dietary records will be performed before the first cooking class to determine habitual dietary intake. The other records will be completed within a week of the week-12 visit. Diet quality will be calculated based on the nutrient intake data. NPCR program will be used to analyze the dietary intakes. HEI-2020 scores will be calculated to measure diet quality and assess alignment with the 2020-2025 DGA.

Dietary Intervention: All participants will attend biweekly cooking classes and food demonstrations at Tucson Village Farm (TVF), a working farm with a teaching kitchen where staff regularly provide direct education to community members related to growing and preparing food to support overall health. During the class, participants in the MyPlate (control) group will receive nutrition education in alignment with standard MyPlate (i.e., a nutrition education tool for consumers based on the DGA) messages while participants in the pulse intervention groups will receive that information plus additional content and messages focused on pulses. At each class, a recipe, inspired by MyPlate, will be prepared and tasted by participants.

Participants will receive a 2-week supply of pulses to take home with them at these classes, one week of cooked, and one week of dry pulses. This balance of pulse forms was selected to enhance acceptability and convenience and improve self-stability. Participants in the Pulses1.5 and Pulses3.0 groups will also be asked to complete a weekly consumption log to track their consumption of the pulses that were provided at the cooking class. They will be asked to return this log at the following cooking class.

The Healthy US-Style Dietary Pattern of the DGA recommends 1.5 cup-eq of pulses each week for a 2000-calorie dietary pattern. Pulse doses will be adjusted for a participant's caloric needs. Each participant's caloric needs will be estimated using a mathematical formula. For example, a participant in the Pulses group who needs 1600 calories/day will receive 1 cup-eq of pulses each week and a participant who needs 3000 calories/day will receive 3 cup-eq of pulses each week. Similarly, a participant in the Pulses Plus group who needs 1600 calories/day will receive 2 cup-eq of pulses each week and a participant who needs 3000 calories/day will receive 6 cup-eq of pulses each week.

Any adverse events and/or changes in medication during the study will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old (with no upper age limit)
* Currently consuming less than 1.5 cup-equivalents of pulses per week
* Willing and able to participate in a 12-week dietary intervention focused on increased pulse consumption
* Able to communicate in English and provide written informed consent
* Assessed as suitable to participate in a nutrition intervention by the study dietitian or primary healthcare provider

Exclusion Criteria:

* Individuals already consuming >150 minutes/week of pulse-based dietary programming or otherwise regularly meeting high pulse intake benchmarks at baseline
* Patients with food allergies or intolerances that preclude the consumption of pulses
* Individuals who have not received clearance from their healthcare provider to make significant dietary modifications
* Participants anticipating major changes in dietary habits due to elective surgery, planned relocation, or other lifestyle alterations during the study period (12 weeks)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum LDL cholesterol | baseline, 3 months
  LDL cholesterol will be measured using a standard lipid panel. Blood samples will be collected after an overnight fast and analyzed using standardized laboratory methods. LDL cholesterol will be reported in mg/dL. Minimum Value: 0 mg/dL (theoretically, though not physiologically possible). Maximum value: No absolute upper limit, but values above 190 mg/dL are considered very high and associated with significant cardiovascular risk. Interpretation: <100 mg/dL (Optimal, low risk). ≥190 mg/dL (Very high, significantly increased cardiovascular risk).
Change in serum HbA1c | baseline, 3 months
  HbA1c will be measured using standard laboratory methods (such as high-performance liquid chromatography or immunoassay) to assess the average blood glucose levels over the past 2-3 months. Blood samples will be collected at the specified time points. Minimum Value: 0% (theoretically, though not physiologically possible). Maximum Value: There is no absolute upper limit, but values above 15% are typically associated with severe uncontrolled diabetes. Interpretation: Normal: <5.7%. Diabetes: ≥6.5% (diagnostic threshold for diabetes, confirmed by a repeat test). Diabetes: ≥6.5% (diagnostic threshold for diabetes, confirmed by a repeat test).
Change in Brachial Blood Pressure | baseline, 3 months
  Blood pressure will be measured using a standardized sphygmomanometer or an automated digital device. Measurements will be taken after the patient has been at rest for at least 5 minutes. Both systolic and diastolic blood pressures will be recorded in mmHg at specified time points. Minimum Value: 0 mmHg (theoretically, though not physiologically possible). Maximum Value: There is no absolute upper limit, but very high values, typically above 200/120 mmHg, represent hypertensive crisis and require immediate medical intervention. Interpretation: Normal: Systolic <120mmHg, Diastolic <80mmHg. Hypertension Above: Systolic 130-139mmHg, Diastolic: 80-89mmHg
Change in serum C-Reactive Protein (CRP) | baseline, 3 months
  CRP levels will be measured using a high-sensitivity CRP (hs-CRP) blood test to assess systemic inflammation. A decrease in CRP levels will indicate a reduction in inflammation, potentially reflecting treatment efficacy. Minimum Value: <0.3 mg/L (considered normal). Maximum Value: >10 mg/L (indicative of significant inflammation or infection). Interpretation: <1 mg/L → Low risk of inflammation (cardiovascular risk assessment); >10 mg/L → Suggests acute infection or chronic inflammatory disease.

SECONDARY OUTCOMES:
Change in serum Total Cholesterol | baseline, 3 months
  Total cholesterol levels will be measured through a fasting blood test to assess lipid profile changes. A decrease in total cholesterol levels may indicate improved lipid metabolism and reduced cardiovascular risk. Minimum Value: <125 mg/dL (low cholesterol, potential nutritional deficiencies). Maximum Value: >240 mg/dL (high cholesterol, increased cardiovascular risk)
Change in serum High-Density Lipoprotein Cholesterol (HDL-C) | baseline, 3 months
  HDL-C levels will be measured through a fasting blood test to assess changes in cardioprotective lipid levels. An increase in HDL-C is associated with a reduced risk of cardiovascular disease. Minimum Value: <20 mg/dL (severely low, high cardiovascular risk). Maximum Value: >100 mg/dL (uncommon, but very high levels may have unclear clinical significance)
Change in Serum Triglyceride (TG) | baseline, 3 months
  Triglyceride levels will be measured through a fasting blood test to assess lipid metabolism. A reduction in triglyceride levels may indicate improved cardiovascular and metabolic health. Minimum Value: <30 mg/dL (low levels, potentially associated with malnutrition or metabolic conditions). Minimum Value: <30 mg/dL (low levels, potentially associated with malnutrition or metabolic conditions)
Change in Diet Quality Score (Healthy Eating Index - HEI) | baseline, 3 months
  Diet quality will be assessed using the Healthy Eating Index (HEI-2015 or HEI-2020), which evaluates adherence to the Dietary Guidelines for Americans. A higher HEI score indicates better diet quality, associated with improved health outcomes. Minimum Value: 0 (poor diet quality, minimal adherence to dietary guidelines). Maximum Value: 100 (optimal diet quality, full adherence to dietary guidelines).
Change in Satisfaction with Life Score (SWLS) | baseline, 3 months
  Life satisfaction will be assessed using the Satisfaction With Life Scale (SWLS), a validated 5-item questionnaire measuring subjective well-being. Higher scores indicate greater life satisfaction. Participants will rate each statement on a 7-point Likert scale, with total scores ranging from 5 to 35. Minimum Value: 5 (Extremely dissatisfied with life). Maximum Value: 35 (Extremely satisfied with life).
Change in Satisfaction with Food-related Life Score (SWFoL) | baseline, 3 months
  Food-related life satisfaction will be assessed using the Satisfaction with Food-related Life (SWFoL) Scale, a validated 5-item questionnaire that evaluates an individual's overall satisfaction with food and eating experiences. Each item is rated on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree), with total scores ranging from 5 to 35. Higher scores indicate greater satisfaction with food-related life. Minimum Value: 5 (Very low satisfaction with food-related life). Maximum Value: 35 (Very high satisfaction with food-related life).
Change in Physical Activity | baseline, 3 months
  Physical activity will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). This validated self-report questionnaire captures the number of days and average duration per day participants engaged in vigorous activity, moderate activity, and walking over the past 7 days. It also collects data on sedentary time. Responses are converted to MET-minutes/week using IPAQ scoring protocols. Maximum value: High activity: ≥3,000 MET-min/week. Interpretation: Low activity: <600 MET-min/week, Moderate activity: ≥600 to <3,000 MET-min/week and High activity: ≥3,000 MET-min/week

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tucson Village Farm, Tucson, Arizona
  - University of Arizona, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sievenpiper JL, Kendall CW, Esfahani A, Wong JM, Carleton AJ, Jiang HY, Bazinet RP, Vidgen E, Jenkins DJ. Effect of non-oil-seed pulses on glycaemic control: a systematic review and meta-analysis of randomised controlled experimental trials in people with and without diabetes. Diabetologia. 2009 Aug;52(8):1479-95. doi: 10.1007/s00125-009-1395-7. Epub 2009 Jun 13. PMID 19526214
- [Background] Jayalath VH, de Souza RJ, Sievenpiper JL, Ha V, Chiavaroli L, Mirrahimi A, Di Buono M, Bernstein AM, Leiter LA, Kris-Etherton PM, Vuksan V, Beyene J, Kendall CW, Jenkins DJ. Effect of dietary pulses on blood pressure: a systematic review and meta-analysis of controlled feeding trials. Am J Hypertens. 2014 Jan;27(1):56-64. doi: 10.1093/ajh/hpt155. Epub 2013 Sep 7. PMID 24014659
- [Background] Ha V, Sievenpiper JL, de Souza RJ, Jayalath VH, Mirrahimi A, Agarwal A, Chiavaroli L, Mejia SB, Sacks FM, Di Buono M, Bernstein AM, Leiter LA, Kris-Etherton PM, Vuksan V, Bazinet RP, Josse RG, Beyene J, Kendall CW, Jenkins DJ. Effect of dietary pulse intake on established therapeutic lipid targets for cardiovascular risk reduction: a systematic review and meta-analysis of randomized controlled trials. CMAJ. 2014 May 13;186(8):E252-62. doi: 10.1503/cmaj.131727. Epub 2014 Apr 7. PMID 24710915
- [Background] Ferreira H, Vasconcelos M, Gil AM, Pinto E. Benefits of pulse consumption on metabolism and health: A systematic review of randomized controlled trials. Crit Rev Food Sci Nutr. 2021;61(1):85-96. doi: 10.1080/10408398.2020.1716680. Epub 2020 Jan 25. PMID 31983216
- [Background] Mitchell DC, Marinangeli CPF, Pigat S, Bompola F, Campbell J, Pan Y, Curran JM, Cai DJ, Jaconis SY, Rumney J. Pulse Intake Improves Nutrient Density among US Adult Consumers. Nutrients. 2021 Jul 31;13(8):2668. doi: 10.3390/nu13082668. PMID 34444828